CLINICAL TRIAL: NCT05774327
Title: The Effect of Myofascial Release in Addition to Foot Core Exercises on Lower Extremity Performance in Young Adults With Asymptomatic Flexible Pes Planus
Brief Title: Effect of Myofascial Release in Addition to Foot Core Exercises in Young Adults With Asymptomatic Flexible Pes Planus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Ertuğrul Demirdel, Associate Professor, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-1073
Record Dates: First submitted 2023-03-04; First posted 2023-03-17 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Pes Planus
Keywords: Pes Planus; Foot Core Exercises; Myofascial Release; Foam Rolling
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial: Two parallel treatment groups; participants were randomly allocated to Group 1 [Foam Roller+Foot Core Exercises] and Group 2 [Foot Core Exercises]
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foam Roller+Foot Core Exercises Group (Experimental): Participants in the foam roller+exercise group underwent foam roller application, which is a self-myofascial release method, 2 days a week for 6 weeks in addition to exercises. Medium-hard foam rollers were used in the applications. Foam roller application was performed on thoracolumbar fascia, iliotibial band, hamstring, gastro-soleus, peroneals and plantar fascia for 60 seconds on each region. A metronome was used to determine the rhythm during foam roller application. The rhythm of the metronome was set to 60 beats per minute (60 rpm). When determining the amount of load on the tissue, the participants were told to give the maximum amount of load possible.
  Interventions: Other: Foam Roller; Other: Foot Core Exercises
- Foot Core Exercises Group (Experimental): The foot core exercises in the treatment program for young adults with pes planus were taught to the participants one by one. It was checked that each exercise in the program was performed correctly by the participants. An exercise brochure was prepared and given to all participants so that the participants could learn the exercises better and perform them correctly. The exercise program follow-up of the participants and gradual progression of the difficulty levels were performed by the responsible researcher. The exercises were performed two days a week for six weeks under the supervision of the researcher. On the other days, the exercise program follow-up was checked daily via an online platform.
  Interventions: Other: Foot Core Exercises

INTERVENTIONS:
Other: Foam Roller — Participants will be shown 7 different foot core exercises and will be instructed to do 10 repetitions 3 times a day. For 6 weeks, in addition to foot core exercises, myofascial release will be applied with foam roller 2 days a week. Myofascial release application areas; thoracolumbal fascia, iliotibial band, hamstring, gastro-soleus, peroneal, plantar fascia.
  Other Names: Foot Core Exercises
  Arms: Foam Roller+Foot Core Exercises Group
Other: Foot Core Exercises — Participants will be shown 7 different foot core exercises and will be instructed to do 10 repetitions 3 times a day. Foot core exercises; short foot exercise, toe flexion exercise, heel lift exercise,toe abduction exercise, big toe and other toes extension exercise, front swing exercise, back walking exercises. Participants will do the exercises with the researcher two days a week and the other days follow-up will be provided through the online platform.

SUMMARY:
Pes planus is a foot deformity characterized by a low medial longitudinal arch. It is more common in young adults. With low arch, tension occurs in the plantar fascia. Fascia and soft tissue loading may lead to different musculoskeletal problems such as plantar fasciitis, medial tibial stress syndrome, patellofemoral disorders and back pain. In addition, pes planus can affect individuals' activities of daily living, productivity in occupational settings, and injury risk and performance in sports.

Treatment of pes planus includes strengthening, stretching, taping and orthotics for the foot muscles. Among these applications, strengthening of the foot core muscles is one of the most common and effective methods. By strengthening the foot core muscles, it is aimed to reduce the effect of the kinetic chain. Pes planus is a postural deformity that affects the kinetic and fascial chain, but the treatment program is usually planned regionally. With fascial continuity and fascial conduction, the tension on the plantar fascia in pes planus affects the gastro-soleus, peroneus longus and brevis, hamstring muscles, iliotibial band and thoracolumbar fascia. Stretching of the plantar fascia, which is included in current treatment programs, has only a local effect and thus cannot prevent fascial chain involvement. Myofascial release, one of the methods used to reduce the tension in the fascia, has been used frequently in recent years. Myofascial release is performed with methods such as manual, foam roller and instrument assisted release. Foam roller (cylinder foam) is a practical myofascial release method that can be self-applied by the individual.

In addition to strengthening the intrinsic muscles of the foot in individuals with pes planus, it has been reported that fascial chain involvement should also be taken into consideration due to the tension in the plantar fascia with low arch. This study was planned to investigate the effect of myofascial release methods on lower extremity performance in addition to foot core exercises used effectively in the treatment of pes planus.

DETAILED DESCRIPTION:
This study will be carried out with a Randomized Controlled Prospective Study design. For this study, individuals between the ages of 18-25 years with a fall amount of 10 millimeters or more according to the navicular fall test and flexible pes planus according to Jack's finger lift test will be informed about the study and consent for participation will be obtained. Demographic information of the individuals who accept participation will be collected. This study, 2 randomized groups of young adults with flexible pes planus will be formed and one group will be applied an exercise program including only foot core exercises, while the other group will be applied self myofascial release with foam rollers, which is a myofascial release method, in addition to foot core exercises.

Both the experimental and control groups will receive a program consisting of 7 different foot core exercises, each of which will be progressed gradually for 6 weeks, 3 sets of 10 repetitions per day. A brochure for the exercises will be prepared and given to the participants to do at home. In order to follow up the exercise of the participants, the individuals will be called weekly during this period and exercise follow-up will be performed. The experimental group will also be planned to perform 60 seconds of myofascial release on each tissue on the thoracolumbar fascia, iliotibial band, hamstring, gastro-soleus, peroneals and plantar fascia 2 days a week for 6 weeks with foam roller, which is a self-myofascial release method. The amount of load on the tissue will be determined by instructing the individuals to apply the maximum amount of load possible. At the end of six weeks, the initial evaluations will be performed again on all individuals and the measurement results will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18-25,
* Bilateral navicular drop distance of 10 mm or more,
* Bilateral asymptomatic flexible pes planus,
* Volunteering to participate in the study and being able to continue.

Exclusion Criteria:

* Musculoskeletal disorders other than pes planus,
* Having chronic ankle instability,
* Any lower extremity injury in the last 6 months,
* Receiving a treatment related to pes planus in the last 6 months,
* Use of insoles.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-06-09 (Actual)

PRIMARY OUTCOMES:
Change in Balance | Change from Baseline Y Balance Test Results at 6 weeks.
  The Y balance test is used for balance assessment. A "Y" shaped design is made using three tape measures placed on the ground. After the first tape measure is placed in the anterior (ant) direction, the other two tape measures are placed on the ground in the posteromedial (pm) and posterolateral (pl) directions to form a 135-degree angle. How the test will be performed is clearly explained to the individuals before the test and they are allowed to perform three trials. With the hands on the waist, the fingertip reach in each of the three directions is recorded in centimeters (cm). The maximum distance they can reach in three reaches in each direction is recorded. This process is also repeated while standing on the other limb and recorded. Lower limb length is calculated by measuring the distance between the spina iliaca anterior superior and the medial malleolus with a tape measure. With the results obtained, the normalized reach and the composite reach for both limbs are calculated.

SECONDARY OUTCOMES:
Change in Flexibility | Change from Baseline Sit and Reach Test Results at 6 weeks.
  Flexibility is assessed with the sit and reach test. Individuals are trained on how to perform the sit and reach test using three warm-up trials. All individuals sit with the heels/soles of their feet resting on the box, knees fully extended, and fingertips extended as far as possible in the correct position on the metal slide. Individuals are instructed to reach as far forward as possible by pushing the measurement indicator with their fingertips and to hold the maximum reach for two seconds. Three measurements are recorded and the mean calculated.
Change in Power | Change from Baseline Vertical Jump Test Results at 6 weeks.
  Power will be evaluated by vertical jump test. Individuals are measured in a fully rested state and 3 repetitions of vertical jump with 45 seconds rest interval, the best score is recorded.
Change in Gait | Change from Baseline 10-Meter Walk Test Results at 6 weeks.
  Gait is assessed with the 10-meter walk test. The test is performed at a comfortable walking speed on a 14 m walkway for 10 m walk, start (2 m) and finish (2 m). Measurements are repeated 3 times and the average time is recorded in seconds. Cadence is calculated and recorded during the test.

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba Ulusoy, PT, MSc, Principal Investigator — Ankara Yildirim Beyazıt University; Ertuğrul Demirdel, Assoc.prof., Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yıldırım Beyazıt University, Institute of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sulowska I, Oleksy L, Mika A, Bylina D, Soltan J. The Influence of Plantar Short Foot Muscle Exercises on Foot Posture and Fundamental Movement Patterns in Long-Distance Runners, a Non-Randomized, Non-Blinded Clinical Trial. PLoS One. 2016 Jun 23;11(6):e0157917. doi: 10.1371/journal.pone.0157917. eCollection 2016. PMID 27336689
- [Background] Matias AB, Taddei UT, Duarte M, Sacco IC. Protocol for evaluating the effects of a therapeutic foot exercise program on injury incidence, foot functionality and biomechanics in long-distance runners: a randomized controlled trial. BMC Musculoskelet Disord. 2016 Apr 14;17:160. doi: 10.1186/s12891-016-1016-9. PMID 27075480
- [Background] Unver B, Erdem EU, Akbas E. Effects of Short-Foot Exercises on Foot Posture, Pain, Disability, and Plantar Pressure in Pes Planus. J Sport Rehabil. 2019 Oct 18;29(4):436-440. doi: 10.1123/jsr.2018-0363. Print 2020 May 1. PMID 30860412
- [Background] Moon D, Jung J. Effect of Incorporating Short-Foot Exercises in the Balance Rehabilitation of Flat Foot: A Randomized Controlled Trial. Healthcare (Basel). 2021 Oct 13;9(10):1358. doi: 10.3390/healthcare9101358. PMID 34683038
- [Background] Peacock CA, Krein DD, Silver TA, Sanders GJ, VON Carlowitz KA. An Acute Bout of Self-Myofascial Release in the Form of Foam Rolling Improves Performance Testing. Int J Exerc Sci. 2014 Jul 1;7(3):202-211. doi: 10.70252/DTPM9041. eCollection 2014. PMID 27182404
- [Background] Behm DG, Alizadeh S, Hadjizadeh Anvar S, Mahmoud MMI, Ramsay E, Hanlon C, Cheatham S. Foam Rolling Prescription: A Clinical Commentary. J Strength Cond Res. 2020 Nov;34(11):3301-3308. doi: 10.1519/JSC.0000000000003765. PMID 33105383
- [Background] D'Amico A, Silva K, Gallo J. Time Course of Acute Hip Adduction Range of Motion Changes Following Foam Rolling. Int J Sports Phys Ther. 2021 Apr 1;16(2):431-437. doi: 10.26603/001c.21417. PMID 33842038
- [Background] Park DJ, Lee KS, Park SY. Effects of Two Foot-Ankle Interventions on Foot Structure, Function, and Balance Ability in Obese People with Pes Planus. Healthcare (Basel). 2021 Jun 3;9(6):667. doi: 10.3390/healthcare9060667. PMID 34205155
- [Background] Rose GK, Welton EA, Marshall T. The diagnosis of flat foot in the child. J Bone Joint Surg Br. 1985 Jan;67(1):71-8. doi: 10.1302/0301-620X.67B1.3968149.
- [Background] Shaffer SW, Teyhen DS, Lorenson CL, Warren RL, Koreerat CM, Straseske CA, Childs JD. Y-balance test: a reliability study involving multiple raters. Mil Med. 2013 Nov;178(11):1264-70. doi: 10.7205/MILMED-D-13-00222. PMID 24183777
- [Background] Plisky PJ, Rauh MJ, Kaminski TW, Underwood FB. Star Excursion Balance Test as a predictor of lower extremity injury in high school basketball players. J Orthop Sports Phys Ther. 2006 Dec;36(12):911-9. doi: 10.2519/jospt.2006.2244. PMID 17193868
- [Background] Lai WC, Wang D, Chen JB, Vail J, Rugg CM, Hame SL. Lower Quarter Y-Balance Test Scores and Lower Extremity Injury in NCAA Division I Athletes. Orthop J Sports Med. 2017 Aug 8;5(8):2325967117723666. doi: 10.1177/2325967117723666. eCollection 2017 Aug. PMID 28840153
- [Background] Williams W, Selkow NM. Self-Myofascial Release of the Superficial Back Line Improves Sit-and-Reach Distance. J Sport Rehabil. 2019 Oct 18;29(4):400-404. doi: 10.1123/jsr.2018-0306. Print 2020 May 1. PMID 30860410
- [Background] Gonzalo-Skok O, Sanchez-Sabate J, Izquierdo-Lupon L, Saez de Villarreal E. Influence of force-vector and force application plyometric training in young elite basketball players. Eur J Sport Sci. 2019 Apr;19(3):305-314. doi: 10.1080/17461391.2018.1502357. Epub 2018 Jul 28. PMID 30058461
- [Background] Soulard J, Vaillant J, Balaguier R, Vuillerme N. Spatio-temporal gait parameters obtained from foot-worn inertial sensors are reliable in healthy adults in single- and dual-task conditions. Sci Rep. 2021 May 13;11(1):10229. doi: 10.1038/s41598-021-88794-4. PMID 33986307